CLINICAL TRIAL: NCT04429581
Title: Differences in Fat Mass Estimation Formulas in Physically Active Adult Population and Relation With Skinfold Sums.
Status: Completed | Type: Observational
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Esparza Ros, Director of the International Chair of Kinanthropometry, Universidad Católica San Antonio de Murcia
Other Study IDs: 23/02/2013
Record Dates: First submitted 2020-06-05; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Body Weight Changes; Body Weight
Keywords: Fat mass; Body composition assessement; Health; Antropometry
MeSH Terms: conditions — Body Weight Changes; Body Weight | interventions — Anthropometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Anthropometry

SUMMARY:
The objective of the present study was to analyze the differences between the formulas used to estimate fat mass and to establish the existing relationship with the skinfold sum in anthropometry. A total of 2,458 active subjects participated in the study (mean age: 27.98±7.43 years-old). Basic measurements and skinfolds variables were measured following the guidelines of the International Society for the Advancement in Kinanthropometry (ISAK), and Kerr, Durnin-Womersley, Faulkner and Carter equations were used to assess fat mass. Significative differences were found between all the formulas for the percentage of fat mass and the fat mass in kilograms. The correlations among the skinfolds sums and the different equations were high and significative in all the cases. There were differences between all the formulas used to estimate the fat mass. The six or eight skinfold sums could be a valid and better alternative than the fat mass equations or the BMI to assess the subcutaneous fat mass in physically active adults.

ELIGIBILITY:
Inclusion Criteria:

* To be between 18 and 50 years old and to practice any sport in a regular basis

Exclusion Criteria:

* To have overweight or obesity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The present study was conducted with a sample of 2,458 active subjects (mean age: 27,98±7,43 year-old), 1775 men (mean age: 27,99±7,46 years) and 681 women (mean age: 27,94±7,37 years) from Región de Murcia (Spain)
Sampling Method: Non-Probability Sample
Enrollment: 2458 (Actual)
Dates: Start 2013-02-02 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Fat mass weight | 6 years
  Fat mass weight was assessed with skinfold measurements and different prediction equations. Measured in kilograms
Fat mass percentage | 6 years
  Fat mass percentage was assessed with skinfold measurements and different prediction equations. Measured in percentage of total weight.
Six and eight skinfold sums | 6 years
  Skinfolds were measured with a caliper, using anthropometry technique describes by ISAK

SECONDARY OUTCOMES:
Body Mass Index | 6 years
  Weight and height will be combined to report BMI in kg/m^2
Weight | 6 years
  Measured in kilograms
Height | 6 years
  Measured in meters

IPD SHARING:
Plan to Share IPD: No